CLINICAL TRIAL: NCT00979862
Title: A Phase Ib Study of Cediranib in Combination With Cilengitide in Patients With Recurrent Glioblastoma
Brief Title: Cediranib Maleate and Cilengitide in Treating Patients With Progressive or Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02919; NCI-2012-02919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000654715; 0903 (Other: Adult Brain Tumor Consortium); ABTC-0903 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-12

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — cediranib; Cilengitide

ARMS (1):
- Treatment cediranib maleate, cilengitide) (Experimental): Part A (dose finding): Patients receive cediranib maleate PO once daily on days 1-28 and cilengitide IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Part B (dose expansion): Patients are assigned to 1 of 2 groups according to prior anti-VEGF therapy (yes vs no). Patients in both groups receive cediranib maleate (administered at the safe dose determined in part A) and cilengitide as in part A.
  Interventions: Drug: Cediranib Maleate; Drug: Cilengitide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Drug: Cilengitide — Given IV
  Other Names: EMD 121974; EMD-121974
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of cediranib maleate when given together with cilengitide in treating patients with progressive or recurrent glioblastoma. Cediranib maleate and cilengitide may stop the growth of tumor cells by blocking blood flow to the tumor. Giving cediranib maleate together with cilengitide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of cediranib (cediranib maleate) in combination with cilengitide in patients with recurrent glioblastoma (Part A).

SECONDARY OBJECTIVES:

I. To estimate overall survival. II. To estimate the proportion of radiographic responses in recurrent glioblastoma patients with measurable disease treated with cediranib and cilengitide.

III. To estimate the proportion of patients alive and progression free at 6 months (APF6) in patients with recurrent glioblastoma treated at the safe dose as determined in Part A (Part B).

IV. To explore potential imaging techniques and biomarkers to capture the disease process through treatment.

OUTLINE: This is a dose-escalation study of cediranib maleate. Patients are initially enrolled in the dose-finding portion of the study (part A). Once the safe dose of cediranib maleate is determined, additional patients are enrolled in the dose-expansion portion of the study (part B).

Part A (dose finding): Patients receive cediranib maleate orally (PO) once daily on days 1-28 and cilengitide intravenously (IV) over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Part B (dose expansion): Patients are assigned to 1 of 2 groups according to prior anti-VEGF therapy (yes vs no). Patients in both groups receive cediranib maleate (administered at the safe dose determined in part A) and cilengitide as in part A.

After completion of study therapy, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven glioblastoma which is progressive or recurrent following radiation therapy and/or chemotherapy; patients with previous low grade glioma who progressed after radiotherapy and/or chemotherapy and are biopsied and found to have glioblastoma are eligible
* Patients must have measurable contrast-enhancing progressive or recurrent glioblastoma by magnetic resonance imaging (MRI) imaging within two weeks of starting treatment; patient must be able to tolerate MRIs; computed tomography (CT) scans cannot be substituted for MRIs in this study
* Patients must have recovered from severe toxicity of prior therapy; an interval of at least 3 months must have elapsed since the completion of the most recent course of radiation therapy while at least 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen and at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* White blood cell (WBC) >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) =< 3 × institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 ml/min/1.73m^2 for patients with creatinine levels above institutional normal
* Patients must be able to provide written informed consent
* Patients must have =< 2 recurrences/relapses of their tumor
* Women of childbearing potential must have a negative pregnancy test prior to study entry; cediranib has been shown to terminate fetal development in the rat, as expected for a process dependent on vascular endothelial growth factor (VEGF) signaling; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients may not be breast-feeding a child
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must have a Mini-Mental State Exam score of >= 15
* Patients must not have received prior cilengitide or cediranib therapy for their glioblastoma
* ARM 1 OF THE DOSE EXPANSION COHORT ONLY, the last treatment regimen the patient received must have included anti-VEGF treatment; a period of at least 28 days must have elapsed since the last bevacizumab treatment or a period of at least 21 days since the last short-acting anti-VEGF treatment, before treatment with cediranib/cilengitide can begin ARM 2 OF THE DOSE EXPANSION COHORT ONLY: patients must not have had prior anti-VEGF therapy
* Patients must not be on enzyme-inducing anti-epileptic drugs (EIAED); patients may be on non-enzyme inducing anti-epileptic drugs (NEIAED) or not be taking any anti-epileptic drugs

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients with > 2 prior tumor recurrences/relapses
* Patients receiving concurrent investigational agents; patients may not be receiving any other cancer related investigational agents
* Although the following medications are not contraindicated on this study, each should be used with extreme caution due to potential nephrotoxic effects: vancomycin, amphotericin, pentamidine
* Patients may not be on anti-coagulants (dalteparin, warfarin, etc)
* Patients with a mean QTc > 500 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome or other significant electrocardiogram (ECG) abnormality noted within 14 days of treatment are ineligible
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 7 days apart; however, if the first urinalysis shows no protein, then a repeat urinalysis is NOT required
* Patients with a New York Heart Association classification of III or IV
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib or cilengitide
* Uncontrolled intercurrent illness including, but not limited to, hypertension (blood pressure > 140/90 mm Hg), ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because cediranib is a VEGF inhibitor with known abortifacient effects; breastfeeding should be discontinued if the mother is treated with cediranib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cediranib
* Patients on enzyme-inducing AED (EIAED) are not eligible for treatment on this protocol; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 14 days or more prior to the first dose of cediranib or cilengitide
* Patients whose MRI scan demonstrates intratumoral hemorrhage or peritumoral hemorrhage are not eligible for treatment if deemed significant by the treating physician
* Patients must not have a known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhages in the past
* Patients receiving concurrent VEGF inhibitors are prohibited from participating in this study
* Patients with conditions requiring concurrent drugs or biologics with proarrhythmic potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety profile of cediranib maleate based on the incidence of dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days
  The proportion of patients with serious or life threatening toxicities will be estimated along with 95% confidence intervals.

SECONDARY OUTCOMES:
Change in markers | From baseline to up to 7 days after completion of treatment
  Summarized using descriptive statistics. Statistical graphics such as box plots will be used to present the summary statistics at each time point. The differences before and during treatment will be tested using paired statistics.
Overall survival (OS) | Time from the date of treatment start to the date of death, assessed up to 6 months
  Median time of survival along with 95% confidence interval will be estimated using Kaplan-Meier method.
Progression-free survival | At 6 months
  The probability of 6-month progression-free survival will be estimated using binomial distribution.
Radiographic responses using MRI scan | Up to 6 months
  The probability of the responses will be estimated using binomial distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, Principal Investigator — National Cancer Institute (NCI)
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Adult Brain Tumor Consortium, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin